CLINICAL TRIAL: NCT06470815
Title: Long-Term Follow-up Study of ROADSTER 3 Patients
Brief Title: ROADSTER 3 Extended Follow-up Sub-Study
Status: Terminated | Type: Observational
Why Stopped: The decision to close the study is not related to any safety concerns or newly identified risks to patients.
Sponsor: Silk Road Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: SRM-2024-01
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Carotid Artery Diseases
Keywords: Long-term Follow-up; TCAR
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Standard-risk patients who underwent carotid intervention: Symptomatic or asymptomatic patients with a discrete lesion located in the internal carotid artery (ICA) with or without involvement of the contiguous common carotid artery (CCA), who underwent carotid artery revascularization.
  Interventions: Procedure: Transcarotid Artery Revascularization (TCAR)

INTERVENTIONS:
Procedure: Transcarotid Artery Revascularization (TCAR) — Carotid artery revascularization treated with the FDA-cleared ENROUTE Transcarotid NPS in conjunction with the FDA-approved ENROUTE Transcarotid Stent
  Other Names: Carotid Revascularization; Carotid Artery Stenting

SUMMARY:
The study objective is to evaluate long-term outcomes for participants enrolled in the ROADSTER 3 study and treated with the ENROUTE Transcarotid Stent System (TSS) and ENROUTE Transcarotid Neuroprotection System (NPS).

DETAILED DESCRIPTION:
This is an open label, single arm, multi-center post-market study evaluating long-term outcomes for participants at standard risk for adverse events from carotid endarterectomy who underwent carotid revascularization with the ENROUTE Transcarotid Stent System and the ENROUTE Transcarotid Neuroprotection System in the ROADSTER 3 study.

ELIGIBILITY:
Inclusion Criteria:

* Participants who were enrolled in the ROADSTER 3 study and treated with the ENROUTE TSS and ENROUTE NPS
* Able to provide informed consent

Exclusion Criteria:

* Participants who have exited the ROADSTER 3 study early (i.e., prior to completion of protocol required follow-up) will not participate in the sub-study

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who were enrolled in the ROADSTER 3 study
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Ipsilateral Stroke | 2-years, 3-years, 4-years, and 5-years following the index procedure
  Ipsilateral stroke at 2-years, 3-years, 4-years, and 5-years following the index procedure
Ipsilateral Stroke Mortality | 2-years, 3-years, 4-years, and 5-years following the index procedure
  Ipsilateral stroke mortality at 2-years, 3-years, 4-years, and 5-years following the index procedure
In-stent Restenosis | 2-years and 5-years following the index procedure
  In-stent restenosis ≥70% at 2-years and 5-years

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Dermody, MD, Principal Investigator — Lancaster General Hospital; Jeffrey Jim, MD, Principal Investigator — Abbott Northwestern Minneapolis Heart Institute Foundation; Marc Schermerhorn, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (37):
- United States (37):
  - Valley Vascular Consultants, Huntsville, Alabama
  - HonorHealth, Scottsdale, Arizona
  - Pima Heart & Vascular, Tucson, Arizona
  - University of California, San Diego (UCSD), La Jolla, California
  - Sharp Grossmont, La Mesa, California
  - Morton Plant Hospital, Clearwater, Florida
  - Delray Medical Center, Delray Beach, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - AdventHealth Ocala, Ocala, Florida
  - Northside Vascular, Cumming, Georgia
  - Deaconess Research / Evansville Surgical Associates, Evansville, Indiana
  - Indiana University, Indianapolis, Indiana
  - Acadiana Vascular Clinic / Our Lady Lourdes Heart Hospital, Lafayette, Louisiana
  - Maine Medical Center, Portland, Maine
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - McLaren Heart & Vascular, Bay City, Michigan
  - Corewell Health, Grand Rapids, Michigan
  - Abbott Northwestern, Minneapolis, Minnesota
  - St. Luke's Hospital, Chesterfield, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - New York University, New York, New York
  - The Mount Sinai Hospital, New York, New York
  - University of Rochester, Rochester, New York
  - Bethesda North Hospital, Cincinnati, Ohio
  - Providence Portland Medical Center-Hospital, Portland, Oregon
  - St. Luke's University Hospital, Bethlehem, Pennsylvania
  - UPMC Pinnacle, Harrisburg, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Cardiothoracic and Vascular Surgeons, Austin, Texas
  - Memorial Hermann Southeast, Houston, Texas
  - Houston Methodist Sugarland, Sugarland, Texas
  - Sentara, Norfolk, Virginia
  - Carilion Roanoke Memorial, Roanoke, Virginia
  - Charleston Area Medical Center (CAMC), Charleston, West Virginia